CLINICAL TRIAL: NCT02897388
Title: A Quality Improvement Initiative to Increase Breast Milk Use in a Chinese Neonatal Intensive Care Unit (NICU): a Pilot Study
Brief Title: A Quality Improvement Initiative to Increase Breast Milk Use in a Chinese NICU: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CCCTG1
Record Dates: First submitted 2016-08-31; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Infant, Extremely Premature

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intervention (No Intervention): all very low birth weight infants admitted to the NICU at Fudan University Children's Hospital from January 2015 through March 2015 (which is the period before any intervention started)who meet the enroll criteria
- intervention (Experimental): all very low birth weight infants admitted to the NICU at Fudan University Children's Hospital from April 2015 through June 2016 who meet the enroll criteria. A series of breast milk consume promotion interventions would implemented during this intervention period, which including build local lactation team, set breast milk feeding room, train NICU staff etc.
  Interventions: Other: breast milk consume promotion

INTERVENTIONS:
Other: breast milk consume promotion — (1)Team building: organize a multidisciplinary breast milk consume improvement team；(2) Staff education: one nurse to train in Canada for 1 month as lactation coordinator, lactation consultant from Canada to teach NICU staff for 1 month; (3) Send breastmilk teaching materials for parents to teach mothers about breast milk feeding;(4) allocate an area in the NICU as a breast pumping room with breastfeeding pumps and chairs to support mothers pumping milk and feeding their babies; (5)purchase 10 breast pumps from Medela and establish a loaner program for mothers; (6)provide lactation counseling & promote consistent communication about the benefits of mothers' milk to encourage mothers to provide milk for their infants;(7)Coaching by lactation coordinator and nursing staff
  Arms: intervention

SUMMARY:
To assess the prevalence of breast milk feeding in a NICU in China, to implement a quality improvement program to increase breast milk feeding, and to evaluate its impact.

DETAILED DESCRIPTION:
The benefits of breast milk are well recognized for providing health benefits in early infancy and extending into adulthood, and breast milk feeding is promoted by numerous professional organizations. However, for various reasons, in neonatal intensive care unit in China, most infants are separated from their parents and are fed infant formula exclusively. To address this problem, the investigators propose to carry out a pilot study to assess the prevalence of breast milk feeding in a NICU of a tertiary teaching hospital in China, and then to introduce an intervention program to increase the prevalence of breast milk feeding and to evaluate the impact of this program.

The intervention would include building a nutrition team in the NICU, training of a lactation coordinator and nursing staff by a team from Mount Sinai Hospital, providing parents with education on breast milk feeding, providing access to breast pumps through a lend/lease program and providing a breast pumping room for parents. The investigators will collect data on breast milk feeding, including prevalence and reasons for not breast milk feeding during both the pre-intervention and intervention period. The investigators will also assess the enrolled infants' weight gain from admission to discharge, incidence of nosocomial infection and mortality, and average length of stay in the NICU, to assess the efficacy of the breast milk feeding intervention.

This trial has the potential to dramatically change feeding of infants in Chinese NICUs from exclusive infant formula to breast milk, with potential impacts on nosocomial infection, growth, development and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. all very low birth weight(birthweight ≤ 1500g)infants admitted to the NICU of Children's Hospital of Fudan University
2. informed consent is given

Exclusion Criteria:

1. Presence of breast milk feeding contraindications
2. Severe illness with contraindications for feeding

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 325 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
prevalence of breast milk feeding | up to 18 months
  to compare the breast milk feeding incidence between pre-intervention and intervention period

SECONDARY OUTCOMES:
Necrotizing enterocolitis(NEC) incidence | up to 18 months
  to compare the NEC incidence between pre-intervention and intervention period
Nosocomial infection incidence | up to 18 months
  to compare the nosocomial infection incidence between pre-intervention and intervention period
overall mortality rate | up to 18 months
  to compare the overall mortality rate between pre-intervention and intervention period
time to full feeding | up to 18 months
  to compare the time to full feeding between pre-intervention and intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, Ph.D, Study Chair — Children's Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: No
cause all the patients' data is privacy

REFERENCES:
- [Derived] Zhou Q, Zhang L, Lee SK, Chen C, Hu XJ, Liu C, Cao Y. A Quality Improvement Initiative to Increase Mother's Own Milk Use in a Chinese Neonatal Intensive Care Unit. Breastfeed Med. 2020 Apr;15(4):261-267. doi: 10.1089/bfm.2019.0290. Epub 2020 Mar 4. PMID 32129666